CLINICAL TRIAL: NCT00209443
Title: A Multicentre, Phase 3, Open-Label Study to Assess the Efficacy and Safety of 0.1 mmol/kg Omniscan (Gadodiamide Injection) for Magnetic Resonance Angiography (MRA) of the Aorto-iliac Arteries
Brief Title: A Safety and Efficacy Clinical Study to Evaluate the Narrowing of the Aorto-iliac Arteries While Using Gadodiamide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOV302
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Aorto-iliac Stenosis; Arterial Occlusive Diseases
Keywords: Aorto-iliac Stenosis; Occlusion; Diagnostic Imaging; Omniscan; Magnetic Resonance Angiography; Contrast Media
MeSH Terms: conditions — Arterial Occlusive Diseases; Bites and Stings | interventions — gadodiamide

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (1):
- Gadodiamide Injection (Experimental): All subjects received a single intravenous bolus injection via a power injector of Omniscan (Gadodiamide Injection) at a dose of 0.1 mmol/kg
  Interventions: Drug: Gadodiamide Injection

INTERVENTIONS:
Drug: Gadodiamide Injection
  Other Names: Omniscan

SUMMARY:
Magnetic Resonance Angiography (MRA) is an examination similar to Magnetic Resonance Imaging (MRI) which uses a magnetic field and a contrast medium when needed to visualize blood flow in the arterial vessels throughout the body.

Gadodiamide, a contrast medium, is already approved and is used to image blood vessels by directly injecting it into the vein, but this procedure has not been formally tested to image the aorto-iliac vessels using MR.

The study is designed to determine the presence or absence of a relevant stenosis (ie greater than/equal to 50%) or occlusion in aorto-iliac arteries. Intra-arterial Digital Subtraction Angiography (IADSA) will be used as the standard of truth.

DETAILED DESCRIPTION:
GEHC has decided not to provide this detail

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must be adults with confirmed or suspected aorto-iliac stenosis.
* The subject must have been referred for Digital Subtraction Angiography.

Exclusion Criteria:

* The subject has a known hypersensitivity to either conventional X-ray or gadolinium based MR contrast media including, but not restricted to, the investigational product.
* The subject is lactating.
* The subject is pregnant as defined by a serum or urine beta-HCG pregnancy test obtained within 24 hours before administration of the investigational product.
* The subject received or is scheduled to receive MRI contrast medium within 24 hours prior to or less than 24 hours after administration of the investigational product.
* The subject received or is scheduled to receive X-ray contrast medium within 24 hours prior to or less than 24 hours after administration of the investigational product.
* The subject received an investigational product other than OMNISCAN (gadodiamide) within 30 days prior to OMNISCAN administration or will receive an investigational product within the follow-up period proposed for this study.
* The subject presents any clinically active, serious, life-threatening disease with a life expectancy of less than 6 months.
* The subject has a serum creatinine value of >= 3.5 mg/dL (309.4 µmol/L).
* The subject has previously been included in this study.
* The subject has a contra-indication for MRI according to accepted clinical guidelines.
* The subject has metal implants and/or stents in the aorto-iliac region and/or hip replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2004-09; Primary Completion 2006-02-28 (Actual); Study Completion 2006-02-28 (Actual)

PRIMARY OUTCOMES:
Differences in subject level and vessel level sensitivity and specificity between CE-MRA and TOF-MRA in detecting stenosis,(>50% occlusion) in aorto-iliac arteries. IA-DSA is the truth standard. | 27 hours

SECONDARY OUTCOMES:
Differences in sensitivity, specificity, accuracy, PPV and NPV at subject and/or vessel level between CE-MRA and TOF-MRA in detecting stenosis (50% occlusion) in aorta-iliac arteries; Revascularisation strategies based on CE-MRA, TOF-MRA and IA DSA | 27 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Karl, Study Director — GE Healthcare
Locations (1):
- Amersham Buchler GmbH & Co. KG, Ismaning, Germany